CLINICAL TRIAL: NCT06566885
Title: Multicentre, Single Arm, Non-interventional, Observational, Prospective Study to Assess Demographic Characteristics, Burden of Disease and Short-term Patient Reported Outcomes on Symptom Relief in Severe Asthma Patients Aged Older Than 12 Qualifying for Treatment With Tezepelumab in Russia
Brief Title: Real-world Study Assessing Efficacy of TezepeLumaB in Patients With Severe Asthma Regardless of Phenotype in Russia
Acronym: ELBRUS
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5180R00029
Record Dates: First submitted 2024-06-17; First posted 2024-08-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Severe Asthma
Keywords: tezepelumab; severe asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ELBRUS is a 12-month (52-week), multi-centre, prospective, non-comparative and non-interventional (observational), post-reimbursement real-world evidence study that will assess patient-reported outcomes after tezepelumab treatment initiation in participants with severe asthma in Russia.

DETAILED DESCRIPTION:
This is a multi-centre, retrospective-prospective, non-comparative and non-interventional (observational) cohort study involving primary and secondary data collection within real-world settings of participants who initiate tezepelumab for treatment of severe uncontrolled asthma. Participants of the study will be the patients eligible for tezepelumab treatment based on the assessment in accordance with the approved product Summary of Product Characteristics (SmPC) in Russia. The administration of tezepelumab will be independent of this study (i.e., a decision of tezepelumab initiation is based on the physician's choice and regulatory and clinical features, not on recruitment/participation in the study). Tezepelumab is indicated as an add-on maintenance treatment for severe asthma, therefore, patients will continue background asthma therapy throughout the study, irrespective of their decision to participate in this study or not.

Approximately 110 eligible participants of both sexes, aged 12 years or older will be treated with tezepelumab available in the market and according to the Russian reimbursement policies in approximately 20 sites. In eligible participants who agree to take part in the study, the enrolment date is defined as the date of informed consent or assent. After enrolment and evaluation of inclusion/exclusion criteria, study participants will commence tezepelumab treatment as per the physician's decision and following the local product SmPC. The index date is defined as the date when participants have received the first dose of tezepelumab. The enrolment period is the period between enrolment date and index date. Additionally, participants may be enrolled in this study up to 4 weeks after the first dose of tezepelumab, but no longer, to avoid responder bias.

Participants will be followed for a maximum period of 52 weeks after index date, irrespective of treatment discontinuation. Patient-reported outcomes - the primary endpoint (ACQ-5) and SNOT-22 will be retrospectively collected during enrolment for all patients (i.e. the most recent available values in the 52 weeks prior to index date), and prospectively collected at suggested visits at Weeks 4, 12, 24, and 52 following index date. For patients who initiate treatment after being enrolled into the study the baseline value may be collected prospectively after enrolment before start of treatment.

The baseline period is defined as the 52 weeks prior to the index date. Outcomes of interest, such as severe asthma exacerbations, medication use, and healthcare resource utilization, will be collected during enrolment retrospectively for the baseline period (52 weeks prior to the index date) and then prospectively at Weeks 4, 12, 24, and 52 following index date.

Overall expected duration of the study (from the first patient inclusion to the last patient last visit) is about 2 years or until 110 eligible patients are included to the study and data on these patients are collected, whichever occurs first.

As an observational, this study does not imply any intervention into a routine clinical practice, including choice of treatment modality or additional diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

be eligible for enrolment into this study if all of the following criteria are met:

1. Male or female participants aged 12 years or older at the time of signing the ICF or assent.
2. Prescribed and initiated treatment with tezepelumab according to SmPC and local market reimbursement criteria. A period between treatment initiation and enrolment should be no more than 4 weeks.
3. Diagnosis of asthma established for at least 52 weeks prior to tezepelumab initiation and symptoms confirmed by the Investigator not to be due to alternative diagnoses.
4. Received at least one prescription of medium or high doses of ICS during the 52 weeks prior to tezepelumab initiation, with medium or high doses of ICS defined according to the GINA 2022 (see below Note #1).
5. Use of additional asthma maintenance controller medication(s) in addition to ICS (e.g., LABA, leukotriene receptor inhibitors, theophylline, LAMA, and cromones) for at least 52 weeks prior to tezepelumab initiation. The additional maintenance controller medication may be contained in a combination product (e.g., ICS/LABA).
6. Documented history of at least 2 severe asthma exacerbations during the 52 weeks prior to tezepelumab initiation. For participants receiving prior biologic drugs for ≥ 8 months, at least 1 severe exacerbation must have occurred on prior biologic treatment. Participants are excluded if, in the opinion of the Investigator, prior biologic treatment had provided significant clinical benefit in the past 52 weeks, despite the participant experiencing ≥ 2 severe exacerbations during 52 weeks prior to tezepelumab initiation.
7. Individuals with ACQ-5 score ≥ 1.5 (indicating inadequate asthma symptom control) at enrolment or up to 12 weeks before enrolment.
8. Currently receive care from specialist physicians (e.g., pulmonologists and/or allergists) at the Investigator's or sub-Investigator's site.
9. Provision of signed and dated written informed consent, including assent (informed consent for participants under 18 years old).
10. Participants are able to read, understand and complete the questionnaires required by the protocol.

Exclusion Criteria:

1. Any contraindication to tezepelumab as per the approved product SmPC in Russia or in the opinion of the Investigator.
2. Administration of concurrent biologic drug for asthma since the index date, except for stable allergen immunotherapy (defined as a stable dose and regimen at the time of enrolment). Enrolment of patients who were switched from other biologic(s) to tezepelumab is allowed, and an acceptable timeframe since the last prior asthma biologic drug is ≥ 30 days. The number of participants with prior biologic treatment (switching to tezepelumab) should be targeted at 20% or less.
3. Participation in an observational study that might, in the Investigator's opinion, influence the assessment for the current study, or participation in an interventional clinical trial in the last 3 months.
4. Pregnancy or lactation period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants of both sexes, aged 12 years or older with severe uncontrolled asthma despite medium or high doses of ICS, who have commenced/will commence treatment with tezepelumab as determined by their routine clinical care.
  The study population is planned to comprise approximately 110 participants in approximately 20 sites. Eligible patients will be enrolled consecutively at each site to minimize selection bias at each site
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in ACQ-5 score from baseline | 1 year
  time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation. Each question of the Asthma Control Questionnaire-5 is ranged on a 7-point scale from 0 (no impairment) to 6 (maximum impairment). The questions are equally weighted and the ACQ score is the mean of the all questions. The total score of ≥1.5 indicates a high probability that asthma is "poorly controlled", 0-0.75 - that asthma is "well controlled", and 0.75-1.5 is a "grey zone".

SECONDARY OUTCOMES:
1. ACQ-5 score at different points of time | 1 year
  time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation.
  Each question of the Asthma Control Questionnaire-5 is ranged on a 7-point scale from 0 (no impairment) to 6 (maximum impairment). The questions are equally weighted and the ACQ score is the mean of the all questions. The total score of ≥1.5 indicates a high probability that asthma is "poorly controlled", 0-0.75 - that asthma is "well controlled", and 0.75-1.5 is a "grey zone".
2. Proportion of participants with well-controlled asthma | 1 year
  (ACQ-5 score ≤ 0.75) overall during the study and at different points of time [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]
3. Proportion of participants with ACQ-5 response | 1 year
  (reduction of ≥ 0.5 in score from baseline) overall during the study and at different points of time [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]
4. Median time to ACQ-5 response | 1 year
  (reduction of ≥ 0.5 in score from baseline), weeks [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following
8. Pre- and post-bronchodilator forced expiratory volume in 1 second | 2 years
  (FEV1) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]
9. Pre- and post-bronchodilator forced vital capacity | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  (FVC) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]
10. Pre-bronchodilator forced expiratory flow | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  (FEF) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]
11. Changes on pre- and post-bronchodilator FEV1 from baseline | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation.
  Forced expiratory volume in 1 second (FEV1) response is defined as achievement of either a ≥ 5% or ≥ 100 mL improvement from baseline
12. Proportion of pre- and post-bronchodilator FEV1 responders | 1 year
  (defined as participants who achieved either a ≥ 5% or ≥ 100 mL improvement from baseline) overall during the study and at different points of time [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation];
13. FRC | 1 year
  Functional residual capacity (FRC) evaluated by spirometry and/or body plethysmography (if available) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]. Units of measurement: % predicted and L.
14. Annualised rate of severe asthma exacerbations | 2 years
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
15. Proportion of participants with reduced total number of severe asthma exacerbations at Week 52 following tezepelumab initiation compared with baseline | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]:
  a. Proportion of participants with any reduction in severe exacerbations number;
16. Change in annualised rate of severe asthma exacerbations from the baseline period to the follow-up period after tezepelumab initiation | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
17. Proportion of participants with 0, 1, 2, ≥3 severe asthma exacerbations | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
18. Cumulative days of severe asthma exacerbations | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  (calculated in participants who had severe asthma exacerbations at baseline) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
19. Proportion of participants with any SCS use | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  ('systemic' means oral, parenteral CS) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
20. Proportion of participants with any reduction (≥ 25%, ≥ 50%, ≥ 75%, and 100% reduction) from baseline on cumulative SCS dose | during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  (in prednisone equivalent dose) (to be calculated in participants with SCS use at baseline) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
21. Change in median SCS dose from baseline | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  (to be calculated in participants with SCS use at baseline) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
22. Proportion of participants with long-term (>30 consecutive days) SCS use | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  (to be calculated in participants with SCS use at baseline) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
23. Number (proportion) of participants with asthma-related healthcare resource utilisation | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  (by each type) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
24. Annualised rates of asthma-related hospitalisation, emergency calls (or emergency department visits), and unscheduled out-patient visits to a physician | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation];
25. Annualised rates of asthma-related scheduled physician visits or healthcare calls for asthma | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
26. Median overall duration (days) of asthma-related hospitalisations | baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation].
27. Mean and median duration (days) of treatment with tezepelumab | Week 52
  to be calculated in all enrolled participants
28. Median time (days) to tezepelumab discontinuation | Week 52
  to be calculated in participants who discontinued tezepelumab earlier than Week 52 by any reason
29. Proportion of participants discontinued tezepelumab and switched to other biologic drug for asthma treatment and reason(s) | Week 52
8.2 Changes on pre- and post-bronchodilator FVC from baseline | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  Forced Vital Capacity (FVC) (L): both pre-bronchodilator and post-bronchodilator should be recorded. time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
8.3 Changes on pre-bronchodilator FEF from baseline | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  Pre-bronchodilator forced expiratory flow (FEF) 25-75 - the mean speed of flow during forced expiration of from 25% to 75% of the FVC. Measured in L/sec. time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
12.b Proportion of participants with reduced total number of severe asthma exacerbations at Week 52 following tezepelumab initiation compared with baseline | up to 2 years
  [time points to measure: baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]: Proportion of participants with at least 50% reduction in severe exacerbations number;
12.c Proportion of participants with reduced total number of severe asthma exacerbations at Week 52 following tezepelumab initiation compared with baseline | 2 years
  [time points to measure: baseline during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]: c. Proportion of participants who completed 52 weeks of tezepelumab treatment without any severe asthma exacerbation
10.2 RLV | 1 year
  Residual lung volume (RLV) evaluated by spirometry and/or body plethysmography (if available) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]. Units of measurement: % predicted and L.
10.3 TLC | 1 year
  Total lung capacity (TLC) evaluated by spirometry and/or body plethysmography (if available) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation]. Units of measurement: % predicted and L.
5. SNOT-22 questionnaire score | baseline and at Weeks 4, 12, 24, and 52 following tezepelumab initiation
  5. SNOT-22 questionnaire score in patients with comorbid chronic rhinosinusitis with nasal polyps (rhinosinusitis polyposis) at different points of time
6. Proportion of participants with clinically meaningful improvement | baseline and at Weeks 4, 12, 24, and 52 following tezepelumab initiation
  Proportion of participants with clinically meaningful improvement (reduction in SNOT-22 score by ≥ 8.9) overall during the study and at different points of time
7. Median time to SNOT-22 response | baseline and at Weeks 4, 12, 24, and 52 following tezepelumab initiation
  Median time to SNOT-22 response (reduction of ≥8.9 in score from baseline), weeks [time points to measure

OTHER OUTCOMES:
1. Median time from index date to lung function response by FEV1 | 1 year
  (FEV1 response is defined as achievement of either a ≥ 5% or ≥ 100 mL improvement from baseline) [time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation]
2. Proportion of participants with sustained (12 weeks or longer) response by FEV1 | 1 year
  [time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation]
3. Median time from index date to spirometry and/or body plethysmography response | 1 year
  (spirometry and/or body plethysmography response is defined as achievement of a ≥ 5% improvement from baseline) [time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation];
4. Proportion of participants with sustained (12 weeks or longer) spirometry and/or body plethysmography response | 1 year
  [time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation]
5. Proportion of participants with medications for asthma treatment by drug class | 2 years
  [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
6. Cumulative dose of ICS by each ICS medication | 2 years
  (ICS may be contained in a single-component product and a combination product, e.g., ICS/LABA) [time points to measure: during 52 weeks before tezepelumab initiation and up to 52 weeks following tezepelumab initiation]
7. Medication possession ratio (MPR) | Week 52
  total days' supply of a medication in a particular time period, divided by the number of days in the time period
8. A patient's body weight (kg) measured in participants with elevated BMI at enrolment | 1 year
  (≥25 mg/m2) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation];
9. Change in body weight from baseline calculated in participants with elevated BMI at enrolment | 1 year
  (≥25 mg/m2) [time points to measure: baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation].
10. Number and proportion of participants who achieved asthma clinical remission at Week 52 | Week 52
1.2 Median duration of lung function response by FEV1 from index date | 1 year
  time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation
3.2 Median duration of spirometry and/or body plethysmography response from index date (if available) | 1 year
  (spirometry and/or body plethysmography response is defined as achievement of a ≥ 5% improvement from baseline) [time points to measure: baseline and at Weeks 12, 24 and 52 following tezepelumab initiation];
Number and proportion of patients with chronic rhinosinusitis with nasal polyps (CRSwNP) | baseline and at Weeks 4, 12, 24 and 52 following tezepelumab initiation
  Number and proportion of patients with chronic rhinosinusitis with nasal polyps (CRSwNP);
  * Number and proportion of patients with chronic rhinosinusitis without nasal polyps;
  * Number and proportion of patients with CRSwNP with different levels of eosinophils blood count:
    * <150 cells/μl;
    * ≥150 cells/μl;
    * ≥300 cells/μl.
Number and proportion of patients with CRSwNP and presence of biologic therapy prior to tezepelumab initiationor | 1 year
  Number and proportion of patients with CRSwNP and presence of biologic therapy prior to tezepelumab initiationor

CONTACTS AND LOCATIONS:
Locations (15):
- Russia (15):
  - Research Site, Kaliningrad
  - Research Site, Kemerovo
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Nal'chik
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Orenburg
  - Research Site, Petrozavodsk
  - Research Site, Saint Petersburg
  - Research Site, Shelehov
  - Research Site, Stavropol
  - Research Site, Tomsk
  - Research Site, Ulan-Ude
  - Research Site, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/